CLINICAL TRIAL: NCT02064764
Title: Renal Nerve Denervation in Patients With Hypertension and Paroxysmal and Persistent Atrial Fibrillation
Acronym: Symplicity AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Symplicity AF
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Cryoablation only (Active Comparator): Pulmonary vein isolation
  Interventions: Device: Arctic Front Advance™ Cardiac Cryoablation System
- Cryoablation and renal nerve denervation (Experimental): Pulmonary vein isolation plus renal nerve denervation
  Interventions: Device: Symplicity Spyral™ Multi-Electrode Renal Denervation Catheter; Device: Arctic Front Advance™ Cardiac Cryoablation System

INTERVENTIONS:
Device: Symplicity Spyral™ Multi-Electrode Renal Denervation Catheter
  Arms: Cryoablation and renal nerve denervation
Device: Arctic Front Advance™ Cardiac Cryoablation System

SUMMARY:
The purpose of this clinical study is to evaluate the feasibility of performing both renal nerve denervation and pulmonary vein isolation on the same patient with the intent of characterizing both safety and effectiveness in a paroxysmal and persistent atrial fibrillation population with hypertension. To assess safety, the study will measure the occurrence of a composite safety endpoint and, to assess effectiveness, the study will measure freedom of chronic treatment failure through a minimum of six months of follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Drug refractory recurrent symptomatic paroxysmal or persistent atrial fibrillation
* Office-based systolic blood pressure of ≥140 mm Hg based despite treatment with 1 or more antihypertensive medications
* Age 18 years to 80 years old.

Key Exclusion Criteria:

* Renal artery anatomy that is ineligible for treatment including: Lacks at least one renal artery for each kidney with ≥3 mm diameter and minimum treatable length per the Spyral Instructions for Use, Renal artery stenosis (>50%) or renal artery aneurysm in either renal artery, A history of prior renal artery intervention including balloon angioplasty or stenting, Renal artery which contain calcification which does not allow at least four radio frequency ablations to be delivered , Diffuse fibromuscular dysplasia (FMD) or FMD which does not allow at least four radio frequency ablations to be delivered; FMD defined as visible beading of the artery on angiography , Unilateral kidney.
* Estimated Glomerular Filtration Rate of <30 mL/min/1.73m2.
* Pregnant, nursing or planning to be pregnant. (Female participants of childbearing potential must have a negative serum or urine human chorionic gonadotropin (hCG) pregnancy test prior to angiography).
* Currently enrolled or plans to participate in a potentially confounding drug or device trial during the course of this study. Co-enrollment in concurrent studies is allowed when documented pre-approval is obtained from the Medtronic study manager.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Chinitz, MD, Principal Investigator — NYU Langone Health
Locations (10):
- United States (9):
  - Mercy Medical Group-Cardiology, Sacramento, California
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - UPHS-Marquette, Marquette, Michigan
  - NYU Langone Medical Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center Cherry Hill, Seattle, Washington
- Universitätsklinikum des Saarlandes, Homburg, Germany

REFERENCES:
- [Derived] Younis A, Steinberg JS. Renal Denervation for Patients With Atrial Fibrillation. Curr Cardiol Rep. 2021 Jul 16;23(9):126. doi: 10.1007/s11886-021-01558-4. PMID 34269911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on February 6, 2015 and the last subject was enrolled on September 9, 2020
Pre-assignment Details: 28 subjects were exited prior to randomization for not meeting study eligibility criteria. Of the 74 randomized subjects, 3 in the PVI+RDN group were not treated and 1 in the Control group (PVI only) were not treated.
Groups:
- Cryoablation Only: Pulmonary vein isolation
  Arctic Front Advance™ Cardiac Cryoablation System
- Cryoablation and Renal Nerve Denervation: Pulmonary vein isolation plus renal nerve denervation
  Symplicity Spyral™ Multi-Electrode Renal Denervation Catheter
  Arctic Front Advance™ Cardiac Cryoablation System
Period: Overall Study
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Started | 36 | 34
Completed | 30 | 30
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (7.8) | 65.8 (7.8) | 65.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 23 | 16 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not reportable per local laws or regulations | 5 | 4 | 9
  Subject/Physician Chose Not to Provide Information | 2 | 0 | 2
  White | 27 | 28 | 55
  Black or African American | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Hispanic or Latino | 0 | 0 | 0
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52
  Germany | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Each Arm That Experience Safety Composite Events
Description: Characterize the rate of safety composite events, (End stage renal disease, Death, Significant Embolic Event, Renal Artery Perforation or Dissection Requiring Intervention, Vascular Complications, Hospitalization for Hypertensive Crisis, New Renal Artery Stenosis, Cardiac Damage, Pulmonary Vein Stenosis, Atrio-Esophageal Fistula, Arrhythmia, Persistent Phrenic Nerve Palsy), within each of the two study arms and also characterize the difference in the rates between study arms. Each event in the composite has its own time frame, either one month or six months post procedure.
Time Frame: Up to one or six months post procedure depending on the event
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
Participants | 1 | 3
Statistical Analysis 1: Comparison: Cryoablation Only vs Cryoablation and Renal Nerve Denervation; Test type: Other — Log-Rank Test For Comparing Treatment and Control; p = 0.28, Log Rank

2. Primary Outcome: Proportion of Patients With Chronic Treatment Success
Description: Chronic treatment success is freedom from chronic treatment failure. Chronic treatment failure is defined as the occurrence of either a documented episode of AF lasting 2 or more minutes (as measured by an implantable loop recorder) or an intervention for AF.
Time Frame: Minimum of six months
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
Participants | 11 | 10
Statistical Analysis 1: Comparison: Cryoablation Only vs Cryoablation and Renal Nerve Denervation; Test type: Other; p = 0.7348, Log Rank

3. Secondary Outcome: Change in Office Systolic and Diastolic Blood Pressure at 6 Months From Baseline
Description: Compare the difference of office systolic and diastolic blood pressure at 6 months and baseline between study arms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
mmHg
  Office Systolic BP | -11.6 (16.7) | -13.3 (16.8)
  Office Diastolic BP | -5.6 (11.6) | -5.8 (10.0)

4. Secondary Outcome: Difference in Heart Rate at 6 Months and Baseline
Description: Compare the difference in heart rate using the 6 month follow-up measurement and baseline visit measurement. These values will then be compared between study arms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Cryoablation Only: Pulmonary Vein Isolation via Cryoablation
- Cryoablation and Renal Nerve Denervation: PVI via Cryoablation and renal denervation
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
beats per minute | -1.9 (17.3) | 1.8 (16.5)

5. Secondary Outcome: Procedural Measures
Description: Elapsed fluoroscopy time and cryocatheter procedure time between study arms. Renal Denervation Procedure Time and Total Procedural Time will be reported only for the Cryoablation and Renal Denervation group.
Time Frame: Procedure
Population: The analysis population for Renal Denervation Procedure and Total Procedure Time does not include participants from the Cryoablation only group since they did not receive the Renal Artery Denervation Procedure.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
minutes
  Elapsed Fluoroscopy time: number analyzed (Participants) | 36 | 33
  Elapsed Fluoroscopy time | 25.4 (18.9) | 34 (19.8)
  Cryocatheter Procedure Time | 66.2 (25.6) | 68.3 (27.3)
  Renal Artery Denervation Procedure Time: number analyzed (Participants) | 0 | 34
  Renal Artery Denervation Procedure Time |  | 51.2 (16.4)
  Total Procedure Time: number analyzed (Participants) | 0 | 34
  Total Procedure Time |  | 119.5 (35.3)

6. Secondary Outcome: Proportion of Participants With Symptoms at 6 Months Between Study Arms
Description: The endpoints for this objective are presence of the following arrhythmic symptoms as recorded at the 6-month visit through discussion with the patient at the time of the visit:
  * Dizziness
  * Palpitations
  * Rapid heart beat
  * Dyspnea
  * Fatigue
  * Syncope
  * Other
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
Participants
  Dizziness at Baseline | 17 | 11
  Dizziness at 6 months | 6 | 4
  Palpitations at Baseline | 29 | 27
  Palpitations at 6 months | 11 | 9
  Rapid Heart Beat at Baseline | 19 | 18
  Rapid Heart Beat at 6 months | 4 | 6
  Dyspnea at Baseline | 25 | 21
  Dyspnea at 6 months | 6 | 7
  Fatigue at Baseline | 16 | 20
  Fatigue at 6 months | 6 | 8
  Syncope at Baseline | 1 | 1
  Syncope at 6 months | 0 | 0
  Other at Baseline | 13 | 10
  Other at 6 months | 2 | 2

7. Secondary Outcome: Rate of Chronic Treatment Success (Primary Effectiveness Endpoint) for Subjects Off of Class I and III Anti-arrhythmic Drugs Following the Blanking Period.
Description: Compare the rate of chronic treatment success (primary effectiveness endpoint) between study arms for subjects off of Class I and III anti-arrhythmic drugs following the blanking period.
Time Frame: 6 months
Population: If a subject has not used Class I or III anti-arrhythmic drugs at all following the blanking period, all of their follow-up will be used for this analysis. If a subject has used either Class I or Class III anti-arrhythmic drugs after the blanking period, they will be excluded for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 20 | 24
Participants
  Treatment Failure | 13 | 16
  No Treatment Failure | 7 | 8

8. Secondary Outcome: Percent of Time in AF Burden Over All Follow-up Occurring After the Blanking Period
Description: Compare the Percent of time in AF burden over all follow-up occurring after the blanking period between study arms.
Time Frame: 91 days after the cryoablation procedure date until the last Reveal LINQ device data date.
Measure: Mean (Standard Deviation); unit: Percent of time
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
Percent of time | 2.78 (5.96) | 1.75 (5.35)

9. Post Hoc Outcome: Daily Atrial Arrhythmia Burden From Baseline to End of ILR Recording for Patients Who Had a Mean Burden of Greater Than or Equal to 1 Hour Per Day on the Days They Experienced Atrial Arrhythmia(s)
Description: Calculate the daily atrial arrhythmia burden in hours from baseline to end of the ILR recording. The patients who had a mean burden of 1 or more hours per day on the days they experienced atrial arrhythmias are included in the analysis. From these patients, it is then determined the mean daily atrial arrhythmia burden between groups.
Time Frame: Baseline till end of recording of implantable loop recorder
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 36 | 34
hours | 9.2 (6) | 4.1 (3.5)

10. Post Hoc Outcome: Number of Patients Who Discontinued Class I/III Anti-arrhythmic Drugs
Description: Compare the number of patients who discontinued Class I/III anti-arrhythmic drugs between groups
Time Frame: Baseline till end of follow-up (varies per patient)
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
Number analyzed (Participants) | 22 | 20
Participants | 3 | 9

ADVERSE EVENTS:
Time Frame: From Subject enrollment through study completion. Study completion varied for each patient based upon when the last patient completed their 6 month follow-up visit.
Description: Adverse event that:
  1. led to death
  2. led to serious deterioration in health of the subject, that resulted in
     * life-threatening illness or injury, or
     * permanent impairment of body structure or body function, or
     * in-patient or prolonged hospitalization, or
     * medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to body structure or body function,
  b) led to fetal distress, fetal death or congenital abnormality or birth defect
Arm/Group | Cryoablation Only | Cryoablation and Renal Nerve Denervation
All-Cause Mortality (participants affected / at risk) | 1/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 17/36 | 20/34
Other Adverse Events (participants affected / at risk) | 22/36 | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation Only (N=36) | Cryoablation and Renal Nerve Denervation (N=34)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 9 (10)
Atrial flutter (Cardiac disorders) | 1 (1) | 5 (6)
Atrial tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Puncture site hematoma (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
CHA2DS2-VASc annual stroke risk moderate (Investigations) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (2) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation Only (N=36) | Cryoablation and Renal Nerve Denervation (N=34)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 4 (8)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 2 (3) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric mucosa erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application site erythema (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Implant site haematoma (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site oedema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Phrenic nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Albuminuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 3 (3)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (5)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT02064764/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT02064764/SAP_001.pdf